CLINICAL TRIAL: NCT05205837
Title: A Randomized, Double-blinded, Clinical, Placebo-controlled Trial on the Effects of Therapy With Letrozole and hUman Choriongonadotropin in Male Hypogonadism Induced by Illicit Use of Anabolic Androgenic Steroids on Plasma Reproductive Hormones, Fertility, Withdrawal Symptoms and Myocardial Function - The LUCAS Trial
Brief Title: A Randomized, Double-blinded, Clinical, Placebo-controlled Trial on the Effects of Therapy With Letrozole and hUman Choriongonadotropin in Male Hypogonadism Induced by Illicit Use of Anabolic Androgenic Steroids- The LUCAS Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Caroline Michaela Kistorp, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-20036287; 2020-002612-52 (EudraCT Number)
Record Dates: First submitted 2021-12-10; First posted 2022-01-25 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Hypogonadism; Hypogonadism, Male; Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism; Eunuchism | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Masking: Double (Participant, Investigator) Primary Purpose: Treatment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator - placebo (Placebo Comparator): Intervention: Intramuscular injection - placebo Intervention: Drug: placebo
  Interventions: Drug: Placebo
- Active comparator - treatment (Active Comparator): Intervention: intramuscular injection - hCG Intervention: Drug: Letrozole
  Interventions: Drug: Letrozole 2.5mg, hCG

INTERVENTIONS:
Drug: Letrozole 2.5mg, hCG — Drug -Treatment Intramuscular injektion - Treatment
  Arms: Active comparator - treatment
Drug: Placebo — Drug - Placebo Intramuscular injektion - placebo
  Arms: Active Comparator - placebo

SUMMARY:
The overall objective of this randomized trial is to investigate the effects of treatment of AAS- induced male hypogonadism with combined therapy of letrozole and hCG compared with placebo on reproductive hormone levels, adherence to cessation of AAS use, fertility, cardiac function and quality of life.

DETAILED DESCRIPTION:
A randomized, double-blinded, clinical, placebo-controlled trial enrolling 60 male illicit AAS users with documented AAS-induced hypogonadism after a period > 12 weeks of AAS cessation or a negative urine AAS doping test. Participants will be randomized to two study groups; 24 weeks of treatment with either tablet letrozole (femar®) initial dose of 2.5 mg each day versus tablet placebo. After an initial treatment period of four weeks, intramuscular injections with either hCG, initial dose 1500 IE twice weekly (letrozole group) or isotonic saline twice weekly (placebo group) will be added to therapy if plasma total testosterone level has not increased to target plasma level. Following 24 weeks of therapy, all participants will be observed for another 26 weeks without therapy. The study will have one trial center of recruitment: Department of Endocrinology, Rigshospitalet. Following participation in the study, all participants will be offered referral to an endocrine outpatient clinic if they still display clinical and biochemical signs of male hypogonadism.

A healthy group of 30 young lean eugonadal men, who have never used AAS, will be enrolled as control participants and undergo a screening visit and one visit including same procedures as the screening and randomization visits.

ELIGIBILITY:
Inclusion Criteria:

* • Male sex

  * 18 - 50 years of age
  * Hypogonadism following observational period of a minimum of 12 weeks since AAS discontinuation OR hypogonadism with a urine sample negative for AAS analyses at screening visit: plasma total testosterone ≤ 10 nmol/L AND featuring at least one symptom of male hypogonadism using IIEF in terms of erectile function (IIEF: Q1 - Q5 + Q15; total score < 26) and/or sexual desire (IIEF: Q11 + Q12; total < 7) (1) and/or ADAM questionnaire (YES to three questions other than question 1 and 7) and/or regular use of medical treatment for erectile dysfunction.
  * Motivation for permanent AAS cessation

Exclusion Criteria:

* Established cardiovascular disease

  * Established diabetes of any kind 384
  * Congenital hypogonadal conditions (cryptorchidism, Klinefelter's disease, Kallmann's disease etc.)
  * Previous established hypogonadal conditions due to other causes than illicit use of AAS
  * Current or previous treatment with testosterone on other indication than AAS-induced male hypogonadism
  * Abnormal puberty development (small testes, late or absent pubic hairing, late or absent deepening of voice, etc.)
  * Current or previous pituitary diseases including pituitary tumors
  * Current or previous tumors of the hypothalamus
  * Current or former testicular cancer
  * Current or previous prostate cancer
  * Current or previous breast cancer
  * Other cancers unless complete remission ≥ 5 year
  * Other concomitant disease or makes the patient unsuitable to participate in the study
  * Severely impaired liver function
  * Allergy or hypersensitivity to the active substance (letrozole) or excipients of Letrozol "Accord"® listed in Appendix D
  * Allergy or hypersensitivity to the active substance (hCG) or excipients of Brevactid® listed in Appendix D
  * Established Lapp lactase deficiency or glucose/galactose malabsorption
  * Severe venous phlebitis or current or previous venous thromboembolism
  * Inguinal hernia
  * treatment which according to the investigators' assessment
  * Simultaneous participation in another clinical study
  * Unable to follow treatment instructions in terms of study medication instructions
  * Ongoing criminal behavior in terms of violence or illicit distribution of drugs
  * Currently or in the foreseeable future included in anti-doping programs

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-representation of gender identity
Enrollment: 8 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Change in plasma total testosterone concentration after 24 weeks from baseline | 24 weeks

SECONDARY OUTCOMES:
Number of participants who adhere to AAS cessation after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in total plasma testosterone concentration after 50 weeks from baseline | 50 weeks
Change in plasma total testosterone secretion in response to hCG stimulation after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in basal plasma pituitary gonadotropins, LH and FSH, after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in secretion of plasma pituitary gonadotropins, LH and FSH, in response to GnRH stimulation after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in sperm count after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in sperm motility after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in sperm morphology after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in sperm acrosome reaction after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in sperm DNA fragmenting after 24 and 50 weeks from baseline | 24 and 50 weeks
Change in testicular size assessed using ultrasound after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score IIEF (erectile function and libido) from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score ADAM (hypogonadism) from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score of Major Depression Inventory (MDI) (depression) from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score of (GAD7) (anxiety) from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score of Buss-Perry Aggression scale (BPA) (hostility and aggression) from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score of COBRA (Cognitive complaints in bipolar disorder rating assessment) from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score of the Health Assessment Short Form-36 questionnaire from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score of Body-Q 349 (Perception of own body) from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in questionnaire score of the Inventory of Interpersonal Problems 32-item (IIP32) from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in myocardial function assessed by myocardial flow reserve (mL/min/gr) by Rb-82 PET from baseline and after 24 and 50 weeks | 24 and 50 weeks
Change in cardiac systolic function assessed using left ventricular ejection fraction (LVEF) obtained using echocardiography and 24 and 50 weeks from baseline. | 24 and 50 weeks
Change in cardiac systolic function assessed using left ventricular global longitudinal strain (GLS) obtained using echocardiography and 24 and 50 weeks from baseline. | 24 and 50 weeks
Change in cardiac structure (left ventricular mass) obtained using echocardiography and 24 and 50 weeks from baseline. | 24 and 50 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Michaela Kistorp, professor, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No